A Proof of Concept Study Evaluating the Role of Emerging Ultrasound Technologies in the Assessment and Monitoring of Localised Prostate Cancer in Men on an Active Surveillance Programme

**Participant Information Leaflets and Consent Forms** 



Unique Protocol ID:HullUTH

**ERUP Study**: Participation information sheets and

consent forms

V1 06.12.2021



## Current Research in Ultrasound

# Evaluating the Role of Ultrasound in Prostate Cancer Study (ERUP Study)

# Participation Information sheet – Phase 1

## Why is this research being done?

Prostate cancer can be difficult to detect but improvements in ultrasound technology may help us to identify disease more quickly than we can do now. Micro-ultrasound is a developing technology used in diagnostics to assess the prostate. With support from the local cancer alliance network, the radiology department has recently purchased a new ultrasound machine with this new technology. This machine will enable the team in radiology and urology to look at the prostate for evidence of cancer and determine if this new technology can detect disease at an earlier stage than is possible now.

# Why have I been invited to take part?

You have been referred to urology for investigations of your prostate. The Consultant in charge of your care, or one of the doctors or nurses in your team, have asked us to do an MRI scan of your prostate. This looks at the prostate gland and can highlight areas of change that may indicate the need for biopsy. This research is being undertaken on men who have an MRI of the prostate that we can directly compare with the micro-ultrasound pictures, providing us with a valuable insight into the capabilities of this new technology. The data we collect will help improve diagnosis and biopsy planning for future patients. This is particularly important for men who cannot have MRI scans and to help the NHS cope with the demands for its services.

### What are the benefits for me?

By taking part in this study, you will be helping patients of the future and will be helping Hull remain at the forefront of patient care. The data we collect may not be able to change your treatment but it will help men, like you, who are patients in the future. With your permission, will inform your consultant of anything incidental that we find on the scans as part of this research, and keep in close contact with you throughout.





# How will my scan change if I choose to take part?

You will have a standard MRI scan as requested by your doctor or nurse. After that, we will arrange for you to have an ultrasound scan of your prostate. If you need a biopsy following your MRI, we will arrange to do this research scan at the same time. If you do not need a biopsy, we will arrange a convenient time for you to attend for an ultrasound scan that will be used in this study.

For this study, there will be two different ultrasound machines together in the room rather than one. Your prostate will be scanned using both machines, one after the other. After the scans have been completed we will then continue to undertake the prostate biopsy if needed or we will finish the examination and you will be free to go home.

The scans involve a narrow ultrasound probe being inserted a small way into the rectum. This will be similar to the digital rectal examination that you have had from your doctor or nurse. It will not be painful and we will stop the examination if you feel discomfort. The probe will be moved around a little and pictures of your prostate will be taken. The probe will be removed. A second probe will be inserted and the scan repeated using the new micro-ultrasound technology. Each scan will take no more than 5 minutes to complete.

The initial scan described above will be the same as if this research was not being done. The second examination is being done purely for this research study.

The pictures from the scans will be stored anonymously and will be compared to the MRI scan by independent reviewers, either a radiologist or a specialist sonographer. The outcomes of the reviews will be recorded on a secure, password protected database accessible only to the research team.

We will record the result of your latest prostate serum antigen (PSA) blood test which we access from the hospital electronic record system – this is something we do routinely as knowing your blood tests can be important to relate to the scan pictures we normally look at. We will also record the outcomes of any biopsies you have had taken. This extra information will let us see if there are any ultrasound features of the prostate that match the tissue sample readings the laboratories produce.

# Is there any risk?

There are no known risks of having an ultrasound scan. Ultrasound is a very safe test.



Remarkable people.



# Will this affect my treatment or care?

Being involved in this research will not affect how you are treated or cared for in any way.

## Do I have to take part?

You do not have to take part in this research if you do not want to — it is completely your choice and we will not ask why you have or have not decided to be involved. Not being involved in this research will not affect how you are treated or cared for in any way.

Prior to your MRI you will be contacted by me, Pamela Parker, the lead researcher for this study. I will contact you by 'phone to explain more about our research and to seek your consent to join this study.

## **Travel and Parking**

Travel and parking expenses related to your attendance for this research will be reimbursed by the ultrasound department. Please provide receipts where possible.

# Will my Doctor know I have taken part?

We will let the Consultant in charge of your care know you have taken part as while this will not affect how you are looked after in any way, they are responsible for your care overall. We will also inform your own GP that you have been involved and send them a copy of this information sheet so that they are aware you have been involved.

#### What do I do now

Thank you for considering and taking part in this valuable study. I will contact you prior to your MRI and discuss the study with you. If you are happy to proceed I will make a mutually convenient appointment for the ultrasound scan. This is likely to be the same day and time as your planned prostate biopsy.

One the day of the appointment, there will be an opportunity before you are taken into the scan room to ask any questions you have. If you are happy to take part in the research we will ask you to sign a consent form before you go into the room.

#### Consent

You can change your mind and you can withdraw your consent at any time. If you withdraw from the study you will be asked if we can continue to use your data in accordance with the data protection details that follow in the next section.







## Information about me, Pamela Parker the lead researcher

I am receiving help from the research and development department within the Trust and the University of Hull as part of a PhD study. Hull University Teaching hospitals is sponsoring this research. All data I collect and store is in accordance with the Health Research Association and information can be found via the HRA link: www.hra.nhs.uk/patientdataandresearch

## Your information and data protection

In this research study we will use information from your MRI, ultrasound and biopsy investigations. We will only use information that we need for the research study. We will let very few people know your name or contact details, and only if they really need it for this study.

The data we collect will include your initials and a code number held on the secure hospital server. People will use this information to do the research or to check your records to make sure that the research is being done properly. People who do not need to know who you are will not be able to see your name or contact details. Your data will have a code number instead.

We will keep all information about you safe and secure. Everyone involved in this study will keep your data safe and secure. We will also follow all privacy rules.

Once we have finished the study, we will keep some of the data for a maximum of three years so we can check the results. The data will then be securely deleted. We will write our reports in a way that no-one can work out that you took part in the study.

## What are your choices about how your information is used?

You can stop being part of the study at any time, without giving a reason, but we will keep information about you that we already have.

## Where can you find out more about how your information is used?

You can find out more about how we use your information

### at www.hra.nhs.uk/information-about-patients/

our leaflet available from the urology nurse specialist or from ultrasound, at Castle Hill Hospital,

by asking one of the research team,

by sending an email to me <a href="mailto:pamela.parker6@nhs.net">pamela.parker6@nhs.net</a> or

ResearchDevelopment@nhs.net,

by ringing us on (01482) 623065







Our data protection officer can be contacted via email to <a href="https://example.com/HEYIG@nhs.net">HEYIG@nhs.net</a>





# Participant Consent Form - Phase 1

# Evaluating the Role of Ultrasound in Prostate Cancer Study (ERUP Study)

| Name of Chief Investigator: Pamela Parker | Please confirm agreement<br>to the statements by putting<br>your initials in<br>the boxes below |
|---|---|
| I confirm that I have read and understand the information sheet dated <b>03/11/2021</b> (version <b>2</b> ) for the above study. I have had the opportunity to consider the information, ask questions and have had these answered satisfactorily. | |
| I understand that my participation is voluntary and that I am free to withdraw at any time without giving any reason, without my medical care or legal rights being affected. | |
| I understand that incidental findings may be detected during the scans. I give permission for these to be shared with my consultant | |
| I understand that relevant sections of my medical notes and data collected during the study may be looked at by individuals from regulatory authorities or from the NHS Trust, where it is relevant to my taking part in this research. I give permission for these individuals to have access to my records. | |
| I agree to my consultant being informed of my participation in the study. | |
| I agree to take part in the above study. | |
| Participant Signature Da | ate |
| Name of Participant | |
| Researcher Signature Date | |
| Name of Researcher Pamela Parker | |





### Current Research in Ultrasound

# Evaluating the Role of Ultrasound in Prostate Cancer Study (ERUP Study)

# Participation Information sheet – Phase 2

# Why is this research being done?

Prostate cancer can be difficult to detect but improvements in ultrasound technology may help us to identify disease more quickly than we can do now. Micro-ultrasound is a developing technology used in diagnostics to assess the prostate. The aim of this study is to investigate if micro-ultrasound can be used to help monitor men who have regular review of their prostate and to see if it can detect any changes that may lead to earlier treatment if required.

# Why have I been invited to take part?

You will have previously been investigated for suspected prostate cancer and have had an MRI scan. You may also have had a biopsy of your prostate although not all men do. Your consultant has diagnosed low grade prostate cancer and you are being monitored for any evidence of progression. This is known as active surveillance or watchful waiting. Whilst being monitored you will have regular blood tests and digital rectal examinations. Occasionally you may also be referred for an MRI scan. These routine tests can give us an indication of whether your prostate gland is stable or changing. However, published evidence suggests that micro-ultrasound will be able to add valuable information to the doctors looking after patients being monitored in the future that may lead to earlier treatment than they can currently provide.

# What are the benefits of me joining this research?

This research is being undertaken on men who are being monitored so that we can increase our understanding of the benefits of using micro-ultrasound in the monitoring of prostate cancer. Being able to scan men who are currently being monitored will allow us to compare this new technology with the routine regular tests available. This will provide us with a valuable insight into the capabilities of this new technology. The data we collect will help improve the monitoring of men in the future. By taking part in this trial you will be helping patients of the future and will be helping Hull remain at the forefront of patient care.

The data we collect may not be able to change your treatment but it will help men, like you, who are patients in the future. With your permission, will inform your consultant of anything incidental that we find on the scans as part of this research, and keep in close contact with you throughout.







# How will my monitoring change if I choose to take part?

You will have routine blood tests and digital rectal examinations regularly as part of your prostate monitoring. For this research, you will be invited to have ultrasound scans in addition to the routine tests. The first ultrasound scan will be done in the next few weeks and then every 6-months for the duration of the study. You will be invited to a minimum of 1 and a maximum of 4 scans for this study. We will arrange a convenient time for you to attend for each of the ultrasound scans that will be used in this study.

When you attend for the ultrasound scans, there will be two different ultrasound machines together in the room rather than one. Your prostate will be scanned using both machines, one after the other. After the scans have been completed you will be free to go home.

The scans involve a narrow ultrasound probe being inserted a small way into the rectum. This will be similar to the digital rectal examination that you have had from your doctor or nurse. It will not be painful and we will stop the examination if you feel discomfort. The probe will be moved around a little and pictures of your prostate will be taken. The probe will be removed. A second probe will be inserted and the scan repeated using the new micro-ultrasound technology. Each scan will take no more than 5 minutes to complete.

Both of these scans are being done purely for this research study. They are in addition to your routine care.

The pictures from the scans will be compared to your previous MRI scan by independent reviewers, either a radiologist or a specialist sonographer. If you participated in phase 1 of this study, the pictures will also be compared to the previous ultrasound scans you had taken. The outcomes of the reviews will be recorded on a secure, password protected database accessible only to the research team.

We will record the result of your latest prostate serum antigen (PSA) blood test which we access from the hospital electronic record system – this is something we do routinely as knowing your blood tests can be important to relate to the scan pictures we normally look at. We will also record the outcomes of any biopsies you have previously had taken. This extra information will let us see if there are any ultrasound features of the prostate that match the tissue sample readings the laboratories produce.





# Is there any risk?

There are no known risks of having an ultrasound scan. Ultrasound is a very safe test.

# Will this affect my treatment or care?

Being involved in this research will not affect how you are treated or cared for in any way.

## Do I have to take part?

You do not have to take part in this research if you do not want to — it is completely your choice and we will not ask why you have or have not decided to be involved. Not being involved in this research will not affect how you are treated or cared for in any way.

Once you have been given a diagnosis from the doctor looking after you and agreed a monitoring plan you will be contacted by me, Pamela Parker, the lead researcher for this study. I will contact you by 'phone to explain more about our research and to seek your consent to join this study. Thank you considering this invitation.

## **Travel and Parking**

Travel and parking expenses related to your attendance for this research will be reimbursed by the ultrasound department. Please provide receipts where possible.

## Will my Doctor know I have taken part?

We will let the Consultant in charge of your care know you have taken part as while this will not affect how you are looked after in any way, they are responsible for your care overall. We will also inform your own GP that you have been involved and send them a copy of this information sheet so that they are aware you have been involved.

#### What do I do now?

Thank you for considering and taking part in this valuable study. I will contact you in the next few weeks to discuss the study with you. If you are happy to proceed I will make a mutually convenient appointment for the ultrasound scan.

One the day of the appointment, there will be an opportunity before you are taken into the scan room to ask any questions you have. If you are happy to take part in the research we will ask you to sign a consent form before you go into the room.







#### Consent

You can change your mind and you can withdraw your consent at any time. If you withdraw from the study you will be asked if we can continue to use your data in accordance with the data protection details that follow in the next section.

### Information about me, Pamela Parker the lead researcher

I am receiving help from the research and development department within the Trust and the University of Hull as part of a PhD study. Hull University Teaching hospitals is sponsoring this research. All data I collect and store is in accordance with the Health Research Association and information can be found via the HRA link: www.hra.nhs.uk/patientdataandresearch

# Your information and data protection

In this research study, we will use information from your MRI, ultrasound and biopsy investigations. We will only use information that we need for the research study. We will let very few people know your name or contact details, and only if they really need it for this study.

The data we collect will include your initials and a code number held on the secure hospital server. People will use this information to do the research or to check your records to make sure that the research is being done properly. People who do not need to know who you are will not be able to see your name or contact details. Your data will have a code number instead.

We will keep all information about you safe and secure. Everyone involved in this study will keep your data safe and secure. We will also follow all privacy rules.

Once we have finished the study, we will keep some of the data for a maximum of three years so we can check the results. The data will then be securely deleted. We will write our reports in a way that no-one can work out that you took part in the study.

## What are your choices about how your information is used?

You can stop being part of the study at any time, without giving a reason, but we will keep information about you that we already have.

## Where can you find out more about how your information is used?

You can find out more about how we use your information







at www.hra.nhs.uk/information-about-patients/

our leaflet available from the urology nurse specialist or from ultrasound, at Castle Hill Hospital,

by asking one of the research team,

by sending an email to <a href="mailto:pamela.parker6@nhs.net">pamela.parker6@nhs.net</a> or

ResearchDevelopment@nhs.net,

by ringing us on (01482) 623065

Our data protection officer can be contacted via email to <a href="https://example.com/HEYIG@nhs.net">HEYIG@nhs.net</a>





# Participant Consent Form - Phase 2

# Evaluating the Role of Ultrasound in Prostate Cancer Study (ERUP Study)

| Name of Chief Investigator: Pamela Parker | Please confirm agreement<br>to the statements by putting<br>your initials in<br>the boxes below |
|---|---|
| I confirm that I have read and understand the information sheet dated <b>03/11/2021</b> (ICF version 2) for the above study. I have had the opportunity to consider the information, ask questions and have had these answered satisfactorily. | |
| I understand that my participation is voluntary and that I am free to withdraw at any time without giving any reason, without my medical care or legal rights being affected. | |
| I understand that incidental findings may be detected during the scans. I give permission for these to be shared with my consultant | |
| I understand that relevant sections of my medical notes and data collected during the study may be looked at by individuals from regulatory authorities or from the NHS Trust, where it is relevant to my taking part in this research. I give permission for these individuals to have access to my records. | |
| I agree to my consultant being informed of my participation in the study. | |
| I agree to take part in the above study. | |
| Participant Signature Da | ate |
| Name of Participant | |
| Researcher Signature D | ate |
| Name of Researcher Pamela Parker | |



12



## Current Research in Ultrasound

# Evaluating the Role of Ultrasound in Prostate Cancer Study (ERUP Study)

# Participation Information sheet – Phase 3

## Why is this research being done?

Micro-ultrasound is a developing technology used in diagnostics to assess the prostate. With support from the local cancer alliance network, the radiology department has recently purchased a new ultrasound machine with micro-ultrasound functions. This machine will enable the team in radiology and urology to look at the prostate for early evidence of cancer development. The aim of this study is to investigate if this technology can be used to help monitor men who have regular review of their prostate and to see if it can detect any changes that may lead to earlier treatment if required. This third phase of the study is evaluating the implementation of, and confidence in using, new technology in everyday clinical practice.

# Why have I been invited to take part?

This research is being undertaken on men who are being investigate for suspected prostate cancer, or who are being monitored for signs of prostate cancer progression. We are doing this so that we can increase our understanding of the benefits of using micro-ultrasound in the diagnosis and active surveillance or watchful waiting pathway of prostate cancer.

You have been invited to participate as you currently have an active role within the prostate cancer pathway. You either currently perform transrectal ultrasound imaging of the prostate, interpret MRI prostate imaging or review imaging results as part of the MDT, or a combination of all. The opinions of all health care professionals is invaluable if we are to successfully implement this new technology within the local pathway and help inform the evidence base around prostate imaging.

Being able to scan men who are currently being monitored will allow us to compare this new technology with the routine regular tests available. This will provide us with a valuable insight into the capabilities of this new technology. The data we collect may help improve the diagnosis and monitoring of men in the within the prostate cancer pathway. By taking part in this trial you will be helping patients of the future and will be helping Hull remain at the forefront of patient care.







# What does phase 3 of the research look like and will my role change?

Patients locally, with suspected prostate cancer or those opting for active surveillance or watchful waiting, are being invited into phase 1 or phase 2 of this study. Both phases involve participants having both a standard transrectal ultrasound scan and a second transrectal ultrasound examination with the new micro-ultrasound examination. In your role you will asked to either, perform, interpret or make decisions based on the findings of the new micro-ultrasound. This will be additional work over and above your current routine practice.

To gain an insight and better understanding of how new technology is implemented into everyday clinical practice, your views about the use of micro-ultrasound will be sought and captured using a survey. This survey will be undertaken at the start of the study and repeated between 6 – 12 months later. We are using a survey adapted from the normalisation process theory toolkit. It is important to understand the opportunities and challenges that implementing new technology present so that these can be address as this becomes embedded into patient care. You can find out more about NPT and its aims being following this <a href="link">link</a> <a href="http://www.normalizationprocess.org/what-is-npt/">http://www.normalizationprocess.org/what-is-npt/</a>

The survey will be sent electronically. All responses will be stored on a password protected data base and only accessible to the lead researcher. The responses will be anonymised by the online survey tool prior to being uploaded onto the database by the lead researcher.

# Do I have to take part?

You do not have to take part in this research if you do not want to – it is completely your choice and we will not ask why you have or have not decided to be involved. Not being involved in this research will not affect your current role or clinical practice.

## What do I do now?

Thank you for considering and taking part in this valuable study. I will contact you in the next few weeks to discuss the study with you. If you are happy to proceed I will ensure that you are sent a secure and individual link to the survey. The survey will be sent again in 6-12 months so that any changes in your opinion of this new technology can be captured. A maximum of two surveys will be sent.





### Consent

You can change your mind and you can withdraw your consent at any time. If you withdraw from the study you will be asked if we can continue to use your data in accordance with the data protection details that follow in the next section.

## Information about me, Pamela Parker the lead researcher

I am receiving help from the research and development department within the Trust and the University of Hull as part of a PhD study. Hull University Teaching hospitals is sponsoring this research. All data I collect and store is in accordance with the Health Research Association and information can be found via the HRA link: www.hra.nhs.uk/patientdataandresearch

## Your information and data protection

In this research study we will use information from your survey results to inform how new technology can be implemented in practice. We will only use information that we need for the research study. We will let very few people know your name or contact details, and only if they really need it for this study.

The data we collect will include your initials and a code number held on the secure hospital server. People will use this information to do the research or to check your records to make sure that the research is being done properly. People who do not need to know who you are will not be able to see your name or contact details. Your data will have a code number instead.

We will keep all information about you safe and secure. Everyone involved in this study will keep your data safe and secure. We will also follow all privacy rules.

Once we have finished the study, we will keep some of the data for a maximum of three years so we can check the results. The data will then be securely deleted. We will write our reports in a way that no-one can work out that you took part in the study.

## What are your choices about how your information is used?

You can stop being part of the study at any time, without giving a reason, but we will keep information about you that we already have.

## Where can you find out more about how your information is used?

You can find out more about how we use your information

at www.hra.nhs.uk/information-about-patients/







our leaflet available from the urology nurse specialist or from ultrasound, at Castle Hill Hospital, by asking one of the research team, by sending an email to <a href="mailto:pamela.parker6@nhs.net">pamela.parker6@nhs.net</a> or <a href="mailto:ResearchDevelopment@nhs.net">ResearchDevelopment@nhs.net</a>, by ringing us on (01482) 623065

Our data protection officer can be contacted via email to <a href="https://example.com/HEYIG@nhs.net">HEYIG@nhs.net</a>





# Participant Consent Form - Phase 3

# Evaluating the Role of Ultrasound in Prostate Cancer Study (ERUP Study)

| Name of Chief Investigator: Pamela Parker | Please confirm agreement to the statements by putting your initials in the boxes below |
|---|---|
| I confirm that I have read and understand the information sheet dated <b>03/11/2021</b> (ICF version <b>2</b> ) for the above study. I have had the opportunity to consider the | |
| information, ask questions and have had these answered satisfactorily. | |
| I understand that my participation is voluntary and that I am free to withdraw at any time without giving any reason, without my role or legal rights being affected. | |
| I agree to take part in the above study. | |
| Participant Signature Da | ate |
| Name of Participant | |
| Researcher Signature Da | ate |
| Name of Researcher Pamela Parker | |





### Current Research in Ultrasound

# Evaluating the Role of Ultrasound in Prostate Cancer Study (ERUP Study)

# Participation Information sheet – Phase 4

# Why is this research being done?

Micro-ultrasound is a developing technology used in diagnostics to assess the prostate. With support from the local cancer alliance network, the radiology department was able to purchase a specific machine with micro-ultrasound functions. This machine has enabled the team in radiology and urology to look at the prostate for early evidence of cancer development. The aim of this study has been to investigate if this technology could be used to help monitor men who have regular review of their prostate and to see if it could detect any changes that may lead to earlier treatment if required.

Phase 4 of the study is being undertaken to disseminate and share the results of the clinical trial that has been undertaken. The clinical trial has evaluated the role of multi-parametric and micro-ultrasound in the assessment of the prostate. The study has been undertaken to increase our understanding of the benefits of using micro-ultrasound in the diagnosis and active surveillance or watchful waiting pathway of prostate cancer. We are interested in the opinions and experience of our colleagues working within the field of imaging or prostate cancer care. This study event has been organised so that we can share our results but, also, for us to hear your thoughts and capture these so that we can compare with our own experiences.

The opinions of all health care professionals is invaluable if we are to successfully implement this new technology within the local pathway and help inform the evidence base around prostate imaging.

## Why have I been invited to take part?

You are attending this study event and, therefore, have some background and knowledge of imaging and prostate cancer care. Your feedback will be valuable to us to help us evaluate the usefulness of our trial and its subsequent implementation into every day clinical practice.





## What does phase 4 of the research look like?

Following the presentations and demonstrations today, there will be a question and answer forum. Notes will be taken from this Q&A session and these will be recorded a narrative so that the main themes, barriers and opportunities can be evaluated at a later date. All notes will be taken anonymously and no personal identifiable data will be recorded. No comments recorded will be attributable to any attendee.

This study is being undertaken as part of a PhD thesis with the University of Hull and the Hull Teaching Hospitals Trust.

## Do I have to take part?

You do not have to take part in this research if you do not want to — it is completely your choice and we will not ask why you have or have not decided to be involved. Not being involved in this research will not affect your attendance at this study event. Your comments will not be recorded and will not form part of the narrative review.

### What do I do now?

Thank you for considering and taking part in this valuable study. If you are happy to participate, please sign the accompanying consent form which will be collected by one of the research team. If you would prefer to not be involved, please indicate this on the accompanying form and your preference will be noted.

#### Consent

You can change your mind and you can withdraw your consent at any time. If you withdraw from the study you will be asked if we can continue to use your data in accordance with the data protection details that follow in the next section.

### Information about me, Pamela Parker the lead researcher

I am receiving help from the research and development department within the Trust and the University of Hull as part of a PhD study. Hull University Teaching hospitals is sponsoring this research. All data I collect and store is in accordance with the Health Research Association and information can be found via the HRA link: <a href="https://www.hra.nhs.uk/patientdataandresearch">www.hra.nhs.uk/patientdataandresearch</a>

## Your information and data protection

In this research study, we will use information from the workshop discussions to produce a narrative of main themes related to prostate imaging. We will only







use information that we need for the research study. We will collect a list of participants who consent to being contacted after the workshop. Only the research team will have access to this data and it will be stored on a password-protected database.

The data we collect from the workshop will include notes of discussion but this will not be attributed to individuals or to specific trusts / health care providers. People will use this information to do the research. People who do not need to know who you are will not be able to see your name or contact details. We will keep all information about you safe and secure. Everyone involved in this study will keep your data safe and secure. We will also follow all privacy rules.

Once we have finished the study, we will keep some of the data for a maximum of three years so we can check the results. The data will then be securely deleted. We will write our reports in a way that no-one can work out that you took part in the study.

# What are your choices about how your information is used?

You can stop being part of the study at any time, without giving a reason, but we will keep information about you that we already have.

# Where can you find out more about how your information is used?

You can find out more about how we use your information

## at www.hra.nhs.uk/information-about-patients/

our leaflet available from the urology nurse specialist or from ultrasound, at Castle Hill Hospital,

by asking one of the research team,

by sending an email to <a href="mailto:pamela.parker6@nhs.net">pamela.parker6@nhs.net</a> or

ResearchDevelopment@nhs.net,

by ringing us on (01482) 623065

Our data protection officer can be contacted via email to <a href="https://example.com/HEYIG@nhs.net">HEYIG@nhs.net</a>





# Participant Consent Form - Phase 4

# Evaluating the Role of Ultrasound in Prostate Cancer Study (ERUP Study)

| Name of Chief Investigator: Pamela Parker | Please confirm agreement<br>to the statements by putting<br>your initials in<br>the boxes below |
|---|---|
| I confirm that I have read and understand the information sheet dated <b>03/11/2021</b> (ICF version 2) for the above study. I have had the opportunity to consider the information, ask questions and have had these answered satisfactorily. | |
| I understand that my participation is voluntary and that I am free to withdraw at any time without giving any reason, without my role or legal rights being affected. | |
| I agreed to being contacted after this workshop related to discussions about prostate imaging | |
| I agree to take part in the above study. | |
| I <b>decline</b> to participate in the above study and do not wish for my comments to be recorded | |
| Participant Signature Da | ate |
| Name of Participant | |
| Researcher Signature D | ate |
| Name of Researcher Pamela Parker | |

